CLINICAL TRIAL: NCT04787575
Title: Open-label, Multicentre, Randomized, Parallel Group Study to Assess the Efficacy and Safety of Oxygen-ozone Therapy Plus Oral Antibiotic Therapy in the Treatment of Infections Secondary to Implant of Orthopaedic Devices
Brief Title: Oxygen-ozone Therapy Plus Antibiotic Therapy in the Treatment of Infections Secondary to Implant of Orthopaedic Devices
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Società Scientifica Internazionale di Ossigeno Ozono Terapia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: sOO3T1 Study
Record Dates: First submitted 2021-02-18; First posted 2021-03-08 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Infection
Keywords: Infection; Orthopaedic device
MeSH Terms: conditions — Infections

STUDY DESIGN:
Intervention Model Description: Open-label, multicentre, randomized, parallel group study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Oxygen-ozone therapy plus antibiotic therapy
  Interventions: Procedure: Oxygen-ozone therapy
- Arm B (Other): Antibiotic therapy
  Interventions: Procedure: Oxygen-ozone therapy

INTERVENTIONS:
Procedure: Oxygen-ozone therapy — Oxygen-ozone therapy (group a) will be performed by:
  i) Self-haemoinfusion of 200 cc. with concentrations of 40-50 μg/ml, to be performed two/three times a week, for a time of 6 weeks (for a maximum of 15 sessions); ii) Subcutaneous injections in the perilesional site at the dose of 5 cc. with concentrations of 4 μg,/ml, Cleanse wounds with 100 cc of 5-10 ug ozone gas

SUMMARY:
This is an open-label, multicentre, randomized, parallel group study to evaluate the efficacy of treatment with oxygen-ozone therapy plus oral antibiotic therapy, in comparison with oral antibiotic therapy alone, in the proportion of patients with resolution/improvement of signs and symptoms of infection of the wound (e.g. ulcer, eschar, sore) in the target lesion after 14 days of treatment, in patients with infections secondary to implant of orthopaedic devices.

DETAILED DESCRIPTION:
This will be an open-label, multicentre, randomized, parallel group study. The study plan will include a screening visit (Visit 1, Day -7/-3) in which patients will be screened on the basis of inclusion/exclusion criteria and clinically evaluated.

At the end of the 3-7 days of run-in (Visit 2, Baseline visit, Day 0), patient still eligible will be randomised to one of the two following treatment groups:

1. Oxygen-ozone therapy SIOOT plus antibiotic therapy
2. Antibiotic therapy

Patients in both groups will receive oral antibiotic therapy, which will be prescribed at discretion of the Investigator, based on the results of the colture of the swab collected in the target lesion at the screening visit (and later, if needed) and the associated antibiogram.

Follow-up visits will be performed after 7 days (Visit 3, Day 7), 14 days (Visit 4, Day 14), 28 days (Visit 5, Day 28) and 42 days (Visit 6, End of study, Day 42) from the start of treatment.

A visit window of ± 2 days for the date of Visits 3-5 and of ± 3 days for the date of Visits 6 will be allowed.

Patients prematurely discontinued from the study will perform an 'Early termination visit', in which procedures schedule for Visit 6 (End of study, Day 42) will be performed. In case of premature study discontinuation, the Investigator will duly record the reason for premature withdrawal in the appropriate section of the case report form (eCRF).

Visit 6, or the 'Early termination Visit' will represent the conclusion of patient's participation in the investigation.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent;
2. Male or female aged ≥ 18 years;
3. Patient having undergone surgery for implant of an orthopaedic device in the previous 8 weeks;
4. Presence of at least one (but no more than 3) post-operative wounds in the site of surgery (ulcers, eschars, sores);
5. Presence of at least one symptom (pain, burning, redness and malodour) and at least one sign (erythema, local warmth, swelling, purulent secretion) of infection of at least moderate intensity (score ≥ 2) in the target lesion at the screening visit (Visit 1), to be confirmed again at the baseline visit (Visit 2);
6. Wound area of the target lesion ≤ 100 cm2;
7. Patient with presence at least one pathogen identified in the swab collection in the target lesion, which is amenable to be eradicated with oral antibiotic therapy;
8. In case of multiple wounds (however not more than three), non-target lesions must not overlap with the target one (i.e. the largest one);
9. Patient able to perform the wound self-care at home or care by his/her primary caregiver;
10. Willing to refrain from all non-permitted concomitant medication from the screening visit through to the entire study duration.
11. Female subjects of childbearing potential must have a negative urinary pregnancy test at Screening and must practice a reliable method of contraception throughout the study;
12. Patient able to read and understand the study procedures, the requirements for follow-up visits, willing to provide information at the scheduled evaluations and willing, able and ensuring to comply with the study requirements for the whole study period.

Exclusion Criteria:

1. Wounds without signs of localized infection;
2. Presence of more than four wounds;
3. Presence of one or more wounds with area > 100 cm2;
4. Presence of undermining wounds;
5. Patients with favism, i.e. deficiency of the glucose-6-phosphate dehydrogenase (G6PD) enzyme;
6. Patients with uncontrolled hyperthyroidism;
7. Patients with history of connective tissue disease, e.g., mixed connective tissue disease;
8. Patients with active malignant disease;
9. Patients with other clinically significant diseases, or other major diseases deemed clinically significant by the Investigator or which in the opinion of the Investigator would interfere with the study procedures or study outcome;
10. Patients candidate to any surgery during the overall study duration;
11. Treatment with topical corticosteroids in the previous 4 weeks and/or with systemic corticosteroids in the previous 7 days;
12. Treatment with any hydrating and/or moisturizing cream in the previous 24 hours.
13. Patients on treatment with chemotherapeutic agents, radiation therapy or immunosuppressive therapies;
14. Patients with contraindications to antibiotic therapy;
15. Pregnant, breastfeeding women and female child-bearing potential who are not using a highly effective method of birth control and not willing to use it during the participation to the study;
16. Participation in any clinical research study evaluating another investigational drug or device within 30 days prior to consenting to study entry;
17. Patient unable to understand informed consent or having a high probability of non-compliance with the study procedures and or non-completion of the study according to investigator's judgement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2024-01-24 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Clinical success at Day 14 | 2 week
  Resolution/improvement of signs and symptoms of infection of the wound in the target lesion (i.e. a score ≤ 1 for a maximum of two signs/symptoms) from baseline to Day 14. The following symptoms will be evaluated by patients on a 0-4 point Likert scale (0 = no symptom; 1 = mild symptom; 2 = moderate symptom; 3 = severe symptom; 4 = very severe symptom): pain, burning, redness and malodour.
  The following signs will be evaluated by investigators on a 0-4 point Likert scale (0 = no sign; 1 = mild sign; 2 = moderate sign; 3 = severe sign; 4 = very severe sign): erythema, local warmth, swelling, purulent secretion.

SECONDARY OUTCOMES:
Proportion of patients with clinical success at Day 7, Day 28, and Day 42 | Day 7, Day 28, and Day 42
  Clinical success is defined as resolution/improvement of signs and symptoms of infection of the wound in the target lesion
Time to resolution of all signs and symptoms of infection | 7 weeks
  It is defined as the disappearance (score = 0) of all signs and symptoms of infection of the wound in the target lesion;
Eradication of the pathogen isolated at the screening visit | 7 weeks
  Bacteriological success of the wound in the target lesion at Day 14 (V4) and Day 42 (V6).A bacteriological success is defined as eradication of the pathogen isolated at the screening visit, without superinfection or reinfection with the same pathogen;
Changes from baseline to any post-baseline time-point of the size of the target lesion | 7 weeks
Global assessment of the target lesion at Day 14 and Day 42 | 7 weeks
  Investigators will be requested to score the outcome of the target lesion on a five-grade scale: 1= worsening, 2 = no change, 3 = minimal improvement, 4 = moderate improvement and 5 = good improvement/resolution;
Changes from baseline to any post-baseline time-point in body temperature | 7 weeks
Changes in WBCs count | 7 weeks
  Changes from baseline to Day 14 (V4) and Day 42 (V6) of white blood cells count (a laboratory parameters that is indicative of infection)
Changes in Erythrocyte sedimentation rate | 7 weeks
  Changes from baseline to Day 14 (V4) and Day 42 (V6) of ESR values (a laboratory parameters that is indicative of infection)
Changes in High-sensitivity C-reactive protein | 7 weeks
  Changes from baseline to Day 14 (V4) and Day 42 (V6) of hs-CRP values (a laboratory parameters that is indicative of infection)

OTHER OUTCOMES:
Number of subjects experiencing treatment-emergent adverse events and serious TEAEs | 7 weeks
Number of subjects experiencing local TEAEs in the site of application of the IP | 7 weeks
Changes from baseline to any post-baseline time point in blood pressure | 7 weeks
  Systolic and diastolic blood pressure will be measured at each study visit in sitting position after at least 10 minutes rest
Changes from baseline to any post-baseline time point in heart rate | 7 weeks
  Heart rate will be recorded at each study visit; it will be measured for one minute just prior to the sitting blood pressure measurement.
Changes in haemoglobin values | 7 weeks
  Haematology will be evaluated in the reference local laboratory of each investigational study site at the screening visit (Visit 1, Day -7/-3) and at Visit 4 (Day 14) and Visit 6 (Day 42).
Changes in haematocrit values | 7 weeks
  Haematology will be evaluated in the reference local laboratory of each investigational study site at the screening visit (Visit 1, Day -7/-3) and at Visit 4 (Day 14) and Visit 6 (Day 42).
Changes in red blood cell (RBC) count | 7 weeks
  Haematology will be evaluated in the reference local laboratory of each investigational study site at the screening visit (Visit 1, Day -7/-3) and at Visit 4 (Day 14) and Visit 6 (Day 42).
Changes in platelet count | 7 weeks
  Haematology will be evaluated in the reference local laboratory of each investigational study site at the screening visit (Visit 1, Day -7/-3) and at Visit 4 (Day 14) and Visit 6 (Day 42).
Changes in creatinine values | 7 weeks
  Blood chemistry will be evaluated in the reference local laboratory of each investigational study site at the screening visit (Visit 1, Day -7/-3) and at Visit 4 (Day 14) and Visit 6 (Day 42).
Changes in blood urea nitrogen (BUN) values | 7 weeks
  Blood chemistry will be evaluated in the reference local laboratory of each investigational study site at the screening visit (Visit 1, Day -7/-3) and at Visit 4 (Day 14) and Visit 6 (Day 42).
Changes in glucose values | 7 weeks
  Blood chemistry will be evaluated in the reference local laboratory of each investigational study site at the screening visit (Visit 1, Day -7/-3) and at Visit 4 (Day 14) and Visit 6 (Day 42).
Changes in aspartate aminotransferase (AST) values | 7 weeks
  Blood chemistry will be evaluated in the reference local laboratory of each investigational study site at the screening visit (Visit 1, Day -7/-3) and at Visit 4 (Day 14) and Visit 6 (Day 42).
Changes in alanine aminotransferase (ALT) values | 7 weeks
  Blood chemistry will be evaluated in the reference local laboratory of each investigational study site at the screening visit (Visit 1, Day -7/-3) and at Visit 4 (Day 14) and Visit 6 (Day 42).
Changes in gamma-glutamyl transpeptidase (gamma-GT) values | 7 weeks
  Blood chemistry will be evaluated in the reference local laboratory of each investigational study site at the screening visit (Visit 1, Day -7/-3) and at Visit 4 (Day 14) and Visit 6 (Day 42).
Changes in alkaline phosphatase values | 7 weeks
  Blood chemistry will be evaluated in the reference local laboratory of each investigational study site at the screening visit (Visit 1, Day -7/-3) and at Visit 4 (Day 14) and Visit 6 (Day 42).
Changes in total bilirubin values | 7 weeks
  Blood chemistry will be evaluated in the reference local laboratory of each investigational study site at the screening visit (Visit 1, Day -7/-3) and at Visit 4 (Day 14) and Visit 6 (Day 42).
Changes in sodium values | 7 weeks
  Electrolytes will be evaluated in blood in the reference local laboratory of each investigational study site at the screening visit (Visit 1, Day -7/-3) and at Visit 4 (Day 14) and Visit 6 (Day 42).
Changes in potassium values | 7 weeks
  Electrolytes will be evaluated in blood in the reference local laboratory of each investigational study site at the screening visit (Visit 1, Day -7/-3) and at Visit 4 (Day 14) and Visit 6 (Day 42).
Changes in magnesium values | 7 weeks
  Electrolytes will be evaluated in blood in the reference local laboratory of each investigational study site at the screening visit (Visit 1, Day -7/-3) and at Visit 4 (Day 14) and Visit 6 (Day 42).
Changes in chloride values | 7 weeks
  Electrolytes will be evaluated in blood in the reference local laboratory of each investigational study site at the screening visit (Visit 1, Day -7/-3) and at Visit 4 (Day 14) and Visit 6 (Day 42).
Changes in calcium values | 7 weeks
  Electrolytes will be evaluated in blood in the reference local laboratory of each investigational study site at the screening visit (Visit 1, Day -7/-3) and at Visit 4 (Day 14) and Visit 6 (Day 42).

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Guastafierro, Principal Investigator — PINETA GRANDE HOSPITAL
Locations (6):
- Italy (6):
  - Pineta Grande Hospital, Castel Volturno, Caserta
  - Ospedali Riuniti Torrette, Ancona
  - Università Federico II, Napoli
  - Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone di Palermo, Palermo
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Casa Di Cura Citta' Di Roma, Roma

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cascini F, Franzini M, Andreoli A, Manzotti A, Cadeddu C, Quaranta G, Gentili A, Ricciardi W. Use of oxygen-ozone therapy to improve the effectiveness of antibiotic treatment on infected arthroplasty: protocol for a superiority, open-label, multicentre, randomised, parallel trial. BMJ Open. 2024 Jan 4;14(1):e076739. doi: 10.1136/bmjopen-2023-076739. PMID 38176866